CLINICAL TRIAL: NCT02932202
Title: Women Eating With Interactive Tracking to Gain Healthily Through Term Pregnancy (WEIGHT) Trial
Brief Title: Women Eating With Interactive Tracking to Gain Healthily Through Term Pregnancy Trial
Acronym: WEIGHT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was stopped due to no recruitment
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Scott Graziano, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208756
Record Dates: First submitted 2016-10-10; First posted 2016-10-13 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Pregnancy; Weight Gain
Keywords: Obesity; Pregnancy; Weight Gain
MeSH Terms: conditions — Obesity; Weight Gain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either a medical student assisted program comprising nutritional counselling and web based nutrition tracking methods (i.e., longitudinal nutritional counseling program) or routine follow-up with their primary healthcare specialist (standard of care) using a 1:1 random numbers block allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longitudinal Nutritional Counseling (Experimental): The intervention group will be contacted every 2 weeks by medical students over the phone to provide nutrition counseling and complete a verbal survey. During the phone calls, participants will be asked a series of questions regarding their dietary intake over the course of the last 2 weeks. If any deficiencies are identified, participants will be counseled on those topics
  Interventions: Other: Longitudinal Nutritional Counseling
- Standard Care Counseling (Placebo Comparator): Participants in the control group will receive standard counseling, which includes weights at every visit, and counseling on weight gain goals as perceived necessary by the provider.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Longitudinal Nutritional Counseling
  Arms: Longitudinal Nutritional Counseling
Other: Standard Care
  Arms: Standard Care Counseling

SUMMARY:
Obesity and excessive weight gain in pregnancy have significant associated maternal and fetal complications including gestational diabetes, large for gestational age infants, birth trauma, and stillbirth. The standard of care places the responsibility on the providers during prenatal visits to remind patients of their weight gain goals and provide appropriate counseling. The objective of this study is to evaluate a sustainable medical student-assisted longitudinal program of nutritional counseling and web based nutrition tracking for pregnant women on excessive weight gain during pregnancy and the effects on diet choices and fetal and maternal complications.

DETAILED DESCRIPTION:
Obesity and excessive weight gain in pregnancy have significant associated maternal and fetal complications including gestational diabetes, large for gestational age infants, birth trauma, and stillbirth. The rates of obesity in American adults is 34.9% and the rates of excessive weight gain in pregnancy for all women range from 20-40% with even higher rates seen in the obese. Such high rates are putting mothers and infants at significant risk.· In 2009, the Institute of Medicine outlined clear guidelines for suggested weight gain goals based on pre-pregnancy BMI. Currently only 30-40% of pregnant women are meeting the suggested weight gain goals and the great majority not meeting the goals are gaining excessive weight. However, despite the high prevalence of excessive weight gain, there is little access to insurance covered nutrition counselling. The standard of care places the responsibility on the providers during prenatal visits to remind patients of their weight gain goals and provide appropriate counselling. This can be challenging due to limited time and resources. However, there is good evidence that diet intervention reduces the risk of excessive weight gain by up to 20%. If appropriate nutritional counselling were available to all patients, the rates of excessive weight gain could be significantly impacted and have widespread improvement in pregnancy outcomes. The CDC has made important progress in providing free nutrition resources online to all patients. This study aims to incorporate this free resource with a sustainable ongoing nutrition counselling to impact the rates of excessive weight gain in pregnancy.

The objective of this study is to evaluate a sustainable medical student-assisted longitudinal program of nutritional counseling and web based nutrition tracking for pregnant women on excessive weight gain during pregnancy and the effects on diet choices and fetal and maternal complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy identified less than 15 week 0 days gestational age
* Body mass index greater then or equal to 18

Exclusion Criteria:

* Multiple gestation
* Pre-pregnancy diabetes mellitus
* HIV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Incidence of excessive weight gain | At time of delivery
  To compare the effect of a medical student assisted program of nutritional counseling and web based nutrition tracking to standard of care on the incidence of excessive weight gain in pregnancy based on the Institute of Medicine's guidelines.

SECONDARY OUTCOMES:
Healthy Eating Habits | At time of delivery
  To characterize how a medical student assisted program of nutritional counselling and web based nutrition tracking affects perception of healthy eating habits (e.g servings of dairy, vegetables, protein, healthy meals)
Pregnancy Comorbidity | At time of delivery
  To compare the incidence of maternal outcomes including gestational diabetes, gestational hypertension and preeclampsia for patients receiving nutrition counselling and web based nutrition tracking compared to standard of care controls

CONTACTS AND LOCATIONS:
Overall Officials: Scott Graziano, MD, Principal Investigator — Loyola University

IPD SHARING:
Plan to Share IPD: No
There is no individual participant data.

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Asbee SM, Jenkins TR, Butler JR, White J, Elliot M, Rutledge A. Preventing excessive weight gain during pregnancy through dietary and lifestyle counseling: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):305-12. doi: 10.1097/AOG.0b013e318195baef. PMID 19155899